CLINICAL TRIAL: NCT05040958
Title: Determination of Carotid Atherosclerotic Plaque Load and Neck Circumference in Cranial CT Angiography With Machine Learning Method and Their Relationship With Each Other
Brief Title: Carotid Atherosclerotic Plaque Load and Neck Circumference
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: CAPNET
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Atherosclerosis of Artery; Metabolic Syndrome; Machine Learning
Keywords: Atherosclerosis of Artery; Metabolic Syndrome; Machine Learning
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to establish a deep learning model to automatically detect the presence and scoring of carotid plaques in neck CTA images, and to determine whether this model is compatible with manual interpretations.

DETAILED DESCRIPTION:
Modeling CTA images for carotid artery segments with deep learning method and automatic carotid plaque presence and scoring will be useful and beneficial in clinical practice. The aim of this study is to establish a deep learning model to automatically detect the presence and scoring of carotid plaques in neck CTA images, and to determine whether this model is compatible with manual interpretations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Having cranial CTA withdrawn
* Having blood lipids, HbA1c, blood glucose, AST, ALT measured in 3 months before and 3 months after cranial CTA

Exclusion Criteria:

* Thyroid disease
* Having had neck surgery
* Use of corticosteroids for more than 6 months
* Presence of lymph nodes in the anterior neck
* Hypertrophy of neck muscles

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People having cranial CTA
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-03-28 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Correlation of the machine learning model and manual interpretation | 1 day
  Evaluation of the correlation of the presence of plaque in the carotid segments with manual interpretation in the model obtained by machine learning method

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Han Training and Research Hospital
Locations (1):
- Istanbul MEdeniyet University Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Kadıköy, Istanbul, Turkey (Türkiye)